CLINICAL TRIAL: NCT05743790
Title: The Role of Dietary Intake and Host Genetics in Gut Microbiome Response to Resistant Starch Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1902008575
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: We originally enrolled 196 participants and collected saliva samples for screening to participate in the intervention. Then we enrolled 76 participants in the intervention study. These participants were randomly assigned to one of two parallel arms in the intervention study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: RS2 first (Experimental): Crackers were provided during each of 3 treatment periods in a crossover design. The 3 types of crackers were matched for total carbohydrate content. Treatment period 1 (10 days): After a 3-day ramp up, participants received 120g of crackers/day containing resistant starch type 2 (30g/day) for 7 days; Treatment period 2 (10 days): Participants received control crackers with 100% digestible starch; Treatment period 3 (10 days): After a 3-day ramp up, participants received 120g of crackers/day containing resistant starch type 4 (30g/day) for 7 days. There were 5-day washout periods between the treatment periods.
  Interventions: Dietary Supplement: RS2-control-RS4
- Group B: RS4 first (Experimental): Crackers were provided during each of 3 treatment periods in a crossover design. The 3 types of crackers were matched for total carbohydrate content. Treatment period 1 (10 days): After a 3-day ramp up, participants received 120g of crackers/day containing resistant starch type 4 (30g/day) for 7 days; Treatment period 2 (10 days): Participants received control crackers with 100% digestible starch; Treatment period 3 (10 days): After a 3-day ramp up, participants received 120g of crackers/day containing resistant starch type 2 (30g/day) for 7 days. There were 5-day washout periods between the treatment periods.
  Interventions: Dietary Supplement: RS4-control-RS2

INTERVENTIONS:
Dietary Supplement: RS2-control-RS4 — Group A: Treatment 1 = RS2 (Hi-Maize 260), Treatment 2 = Control (Amioca TF), Treatment 3 = RS4 (Versafibe 1490)
  Arms: Group A: RS2 first
Dietary Supplement: RS4-control-RS2 — Group B: Treatment 1 = RS4 (Versafibe 1490), Treatment 2 = Control (Amioca TF), Treatment 3 = RS2 (Hi-Maize 260)
  Arms: Group B: RS4 first

SUMMARY:
Resistant starch (RS), a type of dietary fiber, was shown to have beneficial effects on human health through its impact on microbes present in the intestine. However, the effects of RS on the gut microbiota and in turn, on human health, can vary between individuals. Consequently, everyone may not reap the same health benefits by eating high amounts of RS. Factors predicting how an individual's gut microbes as well as the beneficial metabolites produced by these microbes respond to RS supplementation would be helpful in developing precision nutrition approaches that maximize the benefits of dietary fiber intake. The objective of this study was to evaluate candidate predictors of gut microbiota response to RS supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Willing to consume the supplements provided throughout the duration of the study

Exclusion Criteria:

* History of diabetes, prediabetes or impaired glucose tolerance.
* Existing, UNTREATED, thyroid condition.
* Usage of systemic antibiotics (intravenous injection, intramuscular, or oral) within 6 months prior to the study.
* Acute disease at the time of enrollment.
* Chronic, clinically significant pulmonary, cardiovascular, gastrointestinal, hepatic, or renal functional abnormality.
* History of active UNTREATED gastrointestinal disorders or diseases including:

  i. Inflammatory bowel disease (IBD) ii. Ulcerative colitis (mild-moderate-severe) iii. Crohn's disease (mild- moderate-severe) iv. Indeterminate colitis v. Irritable bowel syndrome (IBS) (moderate-severe) vi. Persistent, infectious gastroenteritis, colitis or gastritis vii. Persistent or chronic diarrhea of unknown etiology viii. Clostridium difficile infection (recurrent) ix. Chronic constipation
* Suspected state of immunosuppression or immunodeficiency including HIV.
* History of bariatric surgery.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | 7 weeks
  16S rRNA gene survey of gut microbial communities
Fecal short-chain fatty acid concentration | 7 weeks
  Fecal short-chain fatty acid concentration measurements with ultra-performance liquid chromatography

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States